CLINICAL TRIAL: NCT06277271
Title: E-cigarettes for Harm Reduction in Adults With Opioid Use Disorder
Brief Title: E-cigarettes as a Harm Reduction Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1901611-9
Record Dates: First submitted 2024-01-19; First posted 2024-02-26 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-cigarette (Experimental): Participants will be supplied with an e-cigarette along with a 4-week supply of e-liquid. Participants will receive training on how to use the device and practice puffing with the e-cigarette during the research visit. They will be instructed to self-regulate administration according to their craving and withdrawal symptoms and to refrain from using other nicotine and tobacco products.
  Interventions: Other: E-cigarette

INTERVENTIONS:
Other: E-cigarette — Participants will be supplied with an e-cigarette along with a 4-week supply of e-liquid. Participants will receive training on how to use the device and practice puffing with the e-cigarette during the research visit. They will be instructed to self-regulate administration according to their craving and withdrawal symptoms and to refrain from using other nicotine and tobacco products.

SUMMARY:
E-cigarettes have emerged as an effective strategy for replacing cigarettes among smokers from the general population, but there is a dearth of studies investigating their utility in replacing cigarettes among smokers with opioid use disorder (OUD). This study aims to evaluate the feasibility and acceptability of implementing a cigarette harm reduction intervention involving e-cigarettes in office-based buprenorphine clinics.

DETAILED DESCRIPTION:
Between 84-94% of individuals with opioid use disorder (OUD) smoke cigarettes, a rate six times higher than the general US adult population. Despite the majority of smokers with OUD expressing motivation to quit, cessation rates remain extremely low, even with evidence-based medications. E-cigarettes have emerged as a harm reduction strategy for smokers unable or unwilling to quit. Research on the effectiveness of e-cigarettes for smoking reduction among individuals with OUD on buprenorphine/methadone maintenance treatment is scarce but promising. This study is an open-label single-arm clinical trial testing the use of e-cigarettes as a harm reduction strategy among smokers with OUD on buprenorphine in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥21)
* Report smoking ≥ 5 cigarettes per day for ≥ one year
* Interested in switching to e-cigarettes (self-reported)
* OUD diagnosis (DSM-V)(chart review)
* Currently receiving buprenorphine or other medications for opioid use disorder (MOUD) (chart review)
* Plan to remain on buprenorphine for at least 3 months (duration of the study) (self-reported)
* Have a smartphone with internet access

Exclusion Criteria:

* Use of other tobacco or nicotine products other than cigarettes (≥9 days in the past 30)
* Used nicotine replacement, bupropion or other pharmacotherapies as cessation aids in the past month (bupropion will be allowed for treatment of depression) (self-reported) (3)
* Having a severe medical condition, including decompensated cirrhosis, severe cardiovascular
* disease (myocardial infarction, percutaneous transluminal coronary angioplasty, unstable angina, coronary artery bypass graft, and/or serious arrhythmia in the
* prior 6 months) (chart review)
* Having severe asthma or chronic obstructive pulmonary disease requiring supplemental oxygen or hospitalization in the past 6 months (chart review)
* Being hospitalized for human immunodeficiency virus/acquired immunodeficiency syndromes-related illness in the past 6 months (chart
* review)
* Having a history of seizure disorder (chart review)
* Pregnancy (chart review) or breast-feeding (self-reported) for female participants
* Having current DSM-V criteria for mania, psychosis, or major depressive disorder (chart review)
* Current suicidal ideation or past year suicide attempt (PHQ-9; see protections against risk)
* Being hospitalized for psychiatric reasons in the past year (chart review)
* Being unable to independently read and/or comprehend the consent form or other study materials (unable to read study materials aloud)
* Being unable to read/speak English (inability to read and complete study materials)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Percentage of people who are eligible | Baseline
  Percentage of people who are screened for the study who are eligible and consent to participate in the study
Percentage of consented participants | Through study completion, 1 month follow-up
  Percentage of consented participants will complete the study
Percentage of participants who report using the e-cigarette at least once a day | Week 1 to week 4
  Percentage of participants who report using the e-cigarette at least once a day in weeks 1-4
Percentage of participants with at least one puff of study e-cigarette | Week 1 to week 4
  Percentage of participants with at least one puff of e-cigarette a day in weeks 1-4
Percentage of daily diary completed | Week 1 to week 4
  Percentage of daily diary entries completed

SECONDARY OUTCOMES:
Cigarette dependence measured via the Fagerstrom test for nicotine dependence | Baseline to week 4
  Change in cigarette dependence- baseline vs. week 4
Cigarette demand measured via the cigarette purchase task | Baseline to Week 4
  Change in cigarette demand- baseline vs. week 4
Combustible cigarette smoking | Baseline vs week 4
  Change in average number of cigarettes consumed- baseline vs week 4
Switching to e-cigarettes | week 4
  Percent of participants who switch to e-cigarettes by the end of week 4
Smoking reduction | From baseline to Week 4
  Percent of participants who change their smoking by at least 50%

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No